CLINICAL TRIAL: NCT05548400
Title: Energy and Protein Adequacy of Oral Intake After Ventilator Withdrawal Among Critically Ill Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0070
Record Dates: First submitted 2022-09-06; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Critical Illness; Nutritional Imbalance
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Criticaly ill patients who remained on invasive mechanical ventilation for at least 48 hours.: Criticaly ill patients who remained on invasive mechanical ventilation for at least 48 hours, and dietary followed up after ventilator withdrawal.

SUMMARY:
The aim of this study is to evaluate the adequacy of exclusive oral intake, in terms of energy-protein amount, after extubation in critically ill patients who remained on invasive mechanical ventilation for at least 48 hours.

DETAILED DESCRIPTION:
A prospective observational study. The adequacy of exclusive oral consumption will be assessed in a consecutive sample of critically ill patients after ventilator removal by visual intake scale in 0%, 25%, 50%, 75%, or 100% of principal meals, i.e., lunch and dinner, during seven days after recruitment.

To characterize the study population, general characteristics of patients and their hospital outcomes will be collected: sociodemographic (age, sex, ethnicity, education) and admission clinical data (weight, height, Simplified Acute Physiology Score 3, Nutritional Risk Screening, and Subjective Global Assessment), energy and protein intake within 72 hours after initiation of invasive mechanical ventilation, the underlying disease that led to hospitalization, length of stay in the ICU, length of invasive mechanical ventilation and hospital stay, the incidence of infections after ICU discharge and in-hospital death.

ELIGIBILITY:
Inclusion criteria:

* Adult critically ill patients
* Mechanical ventilation for at least 48 hours and who migrate to exclusively oral feeding within seven days after extubation without receiving complementary parenteral or enteral nutrition.
* Admitted to the ICU in Hospital de Clínicas de Porto Alegre from March 2022 to October 2022.

Exclusion criteria:

* Pregnancy
* Occurrence of major abdominal surgery during ICU stay
* Tracheostomized patients
* Patients unable to start an oral diet after extubation.
* Patients previously included in the study.
* Patients seeking exclusive palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted in the intensive care unit of a general university hospital in southern Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Adequacy of oral intake after extubation on critical ill patients | 7 months
  Oral food intake by an adapted visual intake scale in which the patient or nursing team will indicate intake at 0%, 25%, 50%, or 75 to 100% of principal meals, i.e., lunch and dinner, during seven days after recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana P Antonio, PhD, Principal Investigator — HCPorto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided